CLINICAL TRIAL: NCT03406936
Title: Daily Interruption of Sedation Versus Non Sedation in Mechanically Ventilated Respiratory Failure Patients
Brief Title: Sedation and Ease of Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009917
Record Dates: First submitted 2018-01-13; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Failure; Midazolam Overdose; Chronic Obstructive Pulmonary Disease; Weaning Failure
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily interruption of sedation (Active Comparator): Daily interruption of sedation will be done at 7 am daily by stoppage of midazolam infusion
  Interventions: Drug: Daily interruption of midazolam
- No Sedation (No Intervention): No sedation will be given after initiation of mechanical ventilation

INTERVENTIONS:
Drug: Daily interruption of midazolam — daily at 7 am midazolam infusion will be stopped spontaneous breath trial will be done
  Other Names: sedation interruption
  Arms: Daily interruption of sedation

SUMMARY:
Daily interruption of sedation is one of the modalities which is known to enhance early weaning and separation from mechanical ventilation . Daily sedation interruption is also known to help decreasing incidence of ventilator associated pneumonia. The new modality is no sedation.

DETAILED DESCRIPTION:
there is an increase of incidence of chronic obstructive lung disease associated respiratory failure which necessitates invasive mechanical ventilation. It is well known that one of the bundles for enhanced recovery of such cases is the daily interruption of sedation . Recently studies have demonstrated the feasibility of just using sedation for initiation of mechanical ventilation, then utilization of no sedation technique as a more this offers less side effects .

ELIGIBILITY:
Inclusion Criteria:

* Obstructive lung disease
* Respiratory failure
* Invasive mechanical ventilation

Exclusion Criteria:

* Neurological deficit
* Cognitive dysfunction
* Extensive malignancy
* septic Shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation | first 30 days
  number of days of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt